CLINICAL TRIAL: NCT03736928
Title: A Multicenter, Randomized, Dose-Ranging, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of AbobotulinumtoxinA for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: Safety and Efficacy of AbobotulinumtoxinA for the Treatment of Glabellar Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 43USD1801
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-01

CONDITIONS: Glabellar Frown Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Intramuscular single treatment
  Interventions: Other: placebo
- AbobotulinumtoxinA dose level 1 or 2 (Experimental): Intramuscular single treatment
  Interventions: Biological: AbobotulinumtoxinA dose level 1 or 2
- AbobotulinumtoxinA dose level 3 (Experimental): Intramuscular single treatment
  Interventions: Biological: AbobotulinumtoxinA dose 3
- AbobotulinumtoxinA dose level 4 (Experimental): Intramuscular single treatment
  Interventions: Biological: AbobotulinumtoxinA dose 4

INTERVENTIONS:
Biological: AbobotulinumtoxinA dose level 1 or 2 — Intramuscular; 0.05 mL per injection site; single treatment of glabellar facial lines
  Arms: AbobotulinumtoxinA dose level 1 or 2
Other: placebo — Intramuscular; 0.05 mL per injection site; single treatment of glabellar facial lines
  Arms: Placebo
Biological: AbobotulinumtoxinA dose 3 — Intramuscular; 0.05 mL per injection site; single treatment of glabellar facial lines
  Arms: AbobotulinumtoxinA dose level 3
Biological: AbobotulinumtoxinA dose 4 — Intramuscular; 0.05 mL per injection site; single treatment of glabellar facial lines
  Arms: AbobotulinumtoxinA dose level 4

SUMMARY:
An interventional phase 2 study to evaluate safety and efficacy of AbobotulinumtoxinA treatment for glabellar lines

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe glabellar lines at maximum frown as assessed by the Investigator using a photographic scale
* Moderate to severe glabellar lines at maximum frown as assessed by the subject using a static categorical scale

Exclusion Criteria:

* Botulinum toxin treatment in the face within 9 months prior to study treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Galderma Research Site, Encino, California
  - Galderma Research Site, Manhattan Beach, California
  - Galderma Research Site, Vista, California
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Chicago, Illinois
  - Galderma Research Site, New Orleans, Louisiana
  - Galderma Research Site, New York, New York
  - Galderma Research Site, Chapel Hill, North Carolina
  - Galderma Research Site, Charlotte, North Carolina
  - Galderma Research Site, Mequon, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 401 subjects were randomized, and 399 subjects received study product. Two (2) of the 401 randomized subjects did not receive study product due to hypertension that was identified pre-treatment.
Groups:
- Dose Level 1 AbobotulinumtoxinA; Dose Level 2 AbobotulinumtoxinA: Subjects randomized (4:1) to AbobotulinumtoxinA or placebo
  AbobotulinumtoxinA dose 1/2: treatment of glabellar facial lines
  placebo: treatment of glabellar facial lines
- Dose Level 3 AbobotulinumtoxinA: Subjects randomized (4:1) to dose group 3 AbobotulinumtoxinA or placebo
  placebo: treatment of glabellar facial lines
  AbobotulinumtoxinA dose 3: treatment of glabellar facial lines
- Dose Level 4 AbobotulinumtoxinA: Subjects randomized (4:1) to dose group 4 AbobotulinumtoxinA or placebo
  placebo: treatment of glabellar facial lines
  AbobotulinumtoxinA dose 4: treatment of glabellar facial lines
- Placebo: Subjects randomized to placebo
Period: Overall Study
Arm/Group | Dose Level 1 AbobotulinumtoxinA | Dose Level 2 AbobotulinumtoxinA | Dose Level 3 AbobotulinumtoxinA | Dose Level 4 AbobotulinumtoxinA | Placebo
Started | 80 | 80 | 80 | 81 | 78
Completed | 73 | 78 | 75 | 76 | 67
Not Completed | 7 | 2 | 5 | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 AbobotulinumtoxinA: Subjects randomized (4:1) to dose level 1 AbobotulinumtoxinA or placebo
  AbobotulinumtoxinA dose 1/2: treatment of glabellar facial lines
  placebo: treatment of glabellar facial lines
- Dose Level 2 AbobotulinumtoxinA: Subjects randomized (4:1) to dose level 2 AbobotulinumtoxinA or placebo
  AbobotulinumtoxinA dose 1/2: treatment of glabellar facial lines
  placebo: treatment of glabellar facial lines
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 AbobotulinumtoxinA | Dose Level 2 AbobotulinumtoxinA | Dose Level 3 AbobotulinumtoxinA | Dose Level 4 AbobotulinumtoxinA | Placebo | Total
Number analyzed (Participants) | 80 | 80 | 80 | 81 | 78 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (9.54) | 50.2 (10.33) | 46.3 (11.52) | 48.4 (10.22) | 47.6 (11.5) | 48.4 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 68 | 73 | 68 | 352
  Male | 8 | 9 | 12 | 8 | 10 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 2 | 0 | 5 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2 | 0 | 4
  Black or African American | 4 | 7 | 5 | 6 | 4 | 26
  White | 72 | 67 | 72 | 66 | 71 | 348
  More than one race | 1 | 1 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 2 | 2 | 3 | 1 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 80 | 81 | 78 | 399
Fitzpatrick Skin Type (FST) [Count of Participants; unit: Participants] — FST I: white; very fair; red or blond hair; blue eyes; freckles. always burns, never tans.
  FST II: white; fair; red or blond hair; blue, hazel or green eyes. usually burns, tans with difficulty.
  FST III: cream white; fair with any eye or hair color; very common. sometimes mild burn, gradually tans.
  FST IV: brown; typical Mediterranean Caucasian skin. rarely burns, tans with ease.
  FST V: dark brown; Middle Eastern skin types. very rarely burns, tans very easily.
  FST VI: Skin color - black. Skin Characteristics - never burns, tans very easily.
  Participants
    FST I | 1 | 0 | 1 | 0 | 5 | 7
    FST II | 27 | 21 | 21 | 20 | 17 | 106
    FST III | 32 | 33 | 28 | 28 | 33 | 154
    FST IV | 14 | 12 | 21 | 19 | 19 | 85
    FST V | 4 | 8 | 4 | 8 | 0 | 24
    FST VI | 2 | 6 | 5 | 6 | 4 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Composite Responders at Month 1
Description: composite responder is defined as a subject who achieves a score of 0 or 1 and at least 2 grade improvement on both the Investigator Live Assessment (ILA) and the Subject Self Assessment (SSA)
Time Frame: Month 1 after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 AbobotulinumtoxinA | Dose Level 2 AbobotulinumtoxinA | Dose Level 3 AbobotulinumtoxinA | Dose Level 4 AbobotulinumtoxinA | Placebo
Number analyzed (Participants) | 80 | 80 | 80 | 81 | 78
Participants | 64 | 71 | 72 | 77 | 2

ADVERSE EVENTS:
Time Frame: 36 Weeks
Arm/Group | Dose Level 1 AbobotulinumtoxinA | Dose Level 2 AbobotulinumtoxinA | Dose Level 3 AbobotulinumtoxinA | Dose Level 4 AbobotulinumtoxinA | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/81 | 0/78
Serious Adverse Events (participants affected / at risk) | 1/80 | 3/80 | 0/80 | 1/81 | 0/78
Other Adverse Events (participants affected / at risk) | 3/80 | 1/80 | 1/80 | 4/81 | 2/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 AbobotulinumtoxinA (N=80) | Dose Level 2 AbobotulinumtoxinA (N=80) | Dose Level 3 AbobotulinumtoxinA (N=80) | Dose Level 4 AbobotulinumtoxinA (N=81) | Placebo (N=78)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 AbobotulinumtoxinA (N=80) | Dose Level 2 AbobotulinumtoxinA (N=80) | Dose Level 3 AbobotulinumtoxinA (N=80) | Dose Level 4 AbobotulinumtoxinA (N=81) | Placebo (N=78)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agree not to present or publish any data or reports collected individually or by subgroup of sites prior to full, initial publication based on all data obtained from all sites.

DOCUMENTS (2):
  • Study Protocol (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03736928/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03736928/SAP_001.pdf